CLINICAL TRIAL: NCT00004087
Title: Phase I/II Radioimmunotherapy With High-Dose 90Y-Labeled Humanized MN-14 in Advanced Metastatic Colorectal Cancer and Pancreatic Cancers Using Autologous Peripheral Blood Stem Cell Rescue (PBSCR) to Control Myelotoxicity
Brief Title: Radiolabeled Monoclonal Antibody Therapy Plus Peripheral Stem Cell Transplantation in Treating Patients With Metastatic or Recurrent Colorectal Cancer or Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Garden State Cancer Center at the Center for Molecular Medicine and Immunology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Robert M Sharkey, GSCC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067300; P01CA054425 (NIH); CMMI-C-033-98; NCI-H99-0042; NCI-V99-1571
Record Dates: First submitted 1999-12-10; First posted 2004-04-16 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Colorectal Cancer; Pancreatic Cancer
Keywords: stage IV colon cancer; stage IV pancreatic cancer; recurrent pancreatic cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Pancreatic Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Filgrastim; Peripheral Blood Stem Cell Transplantation; Indium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: filgrastim — as prescribed by physician
Procedure: autologous bone marrow transplantation — 1-2 weeks before treatment
Procedure: peripheral blood stem cell transplantation — 1-2 weeks before treatment
Radiation: indium In 111 monoclonal antibody MN-14 — intravenous infusion over 30 min; single dose
Radiation: yttrium Y 90 monoclonal antibody MN-14 — intravenous infusion over 30 min; single dose

SUMMARY:
RATIONALE: Radiolabeled monoclonal antibodies can locate tumor cells and deliver tumor-killing substances to them without harming normal cells. Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by monoclonal antibody therapy used to kill tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of radiolabeled monoclonal antibody plus peripheral stem cell transplantation in treating patients who have metastatic or recurrent colorectal cancer or pancreatic cancer that has not responded to previous treatment.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose and secondary organ toxicity of high dose yttrium Y 90 monoclonal antibody MN-14 (90Y-hMN-14) plus autologous peripheral blood stem cell rescue in patients with metastatic or recurrent colorectal or pancreatic cancer. II. Compare the tumor to organ dose ratio between 90Y-hMN-14 and iodine 131 monoclonal antibody MN-14 (131I-MN-14) in these patients. III. Determine the antitumor effects with myeloablative doses of 90Y-hMN-14. IV. Evaluate the immunogenicity of 90Y-hMN-14 in these patients.

OUTLINE: This is a dose escalation of yttrium Y 90 monoclonal antibody MN-14 (90Y-hMN-14), multicenter study. Patients are stratified by prior radiotherapy (yes vs no). Patients receive filgrastim (G-CSF) subcutaneously on days -18 to -14 and peripheral blood stem cell (PBSC) collection on days -15 to -13. If an adequate number of CD34+ cells are not harvested, bone marrow is also collected. Patients receive pretherapy imaging with indium In 111 monoclonal antibody MN-14 (IN111-MN-14) IV on days -7 to 0. Patients receive 90Y-hMN-14 for up to 40 minutes on day 0. PBSC are reinfused on days 7 to 14. Patients receive G-CSF SQ until blood counts recover. Cohorts of 3-6 patients receive escalating doses of 90Y-hMN-14 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 3 or 2 of 6 patients experience dose limiting toxicity. Patients are followed at 1-4, 6, 8, 12, and 24 weeks, and then every 6 months thereafter for up to 5 years.

PROJECTED ACCRUAL: A total of 24-30 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven metastatic or recurrent colorectal or pancreatic cancer for which no curative surgery exists Failed at least 1 regimen of standard fluorouracil based chemotherapy for metastatic colorectal cancer or gemcitabine for pancreatic cancer Autologous peripheral blood stem cells (PBSC) or bone marrow available Diffuse bone marrow involvement allowed if: Autologous bone marrow or PBSC with no greater than 5% tumor involvement available Tumor site at least 2.0 cm in diameter confirmed by pretherapy indium In 111 monoclonal antibody MN-14 imaging and CT scan

PATIENT CHARACTERISTICS: Age: 18 to 80 Performance status: Karnofsky 70-100% ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: WBC at least 3,000/mm3 Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 2 mg/dL SGOT no greater than 2.0 times upper limit of normal (ULN) Renal: Creatinine no greater than ULN Other: No severe anorexia, nausea, or vomiting No concurrent significant medical complications that would preclude compliance Not pregnant Fertile patients must use effective contraception during and for 3 months after study No allergy to 90Y-hMN-14

PRIOR CONCURRENT THERAPY: Biologic therapy: Prior murine monoclonal antibody allowed Chemotherapy: No prior irinotecan At least 4 weeks since prior chemotherapy and recovered (8 weeks since nitrosourea, mitomycin or 90Y-hMN-14) Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy to index lesion and recovered No prior radiotherapy to greater than 25% of red marrow (pelvic field radiation as adjuvant therapy for rectal cancer allowed) No prior radiotherapy to maximum tolerated dose to any critical organ (e.g., lung, liver, or kidney) Surgery: At least 4 weeks since major surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 1997-03; Primary Completion 2001-05 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jack D. Burton, MD, Study Chair — Garden State Cancer Center at the Center for Molecular Medicine and Immunology
Locations (3):
- United States (3):
  - Garden State Cancer Center, Belleville, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania